CLINICAL TRIAL: NCT02137161
Title: The Reggio Emilia Study on Bromfenac for Patients With PseudoEXfoliation Syndrome Undergoing Cataract Surgery: the REPEX Study
Brief Title: Bromfenac to Reduce Inflammation in Patients With Pseudoexfoliation Syndrome After Cataract Surgery
Acronym: REPEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-002066-39
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2014-10

CONDITIONS: Cataract; Pseudoexfoliation Syndrome
MeSH Terms: conditions — Cataract; Exfoliation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone+Tobramycin eye drop (Active Comparator): An antibiotic and steroid eye drop association will be given starting the day after the surgery for two weeks, dosed QID for the first week and BID for the second week, to 31 patients.
  Interventions: Drug: Dexamethasone+Tobramycin eye drop
- Bromfenac (Experimental): Bromfenac eye drops (BID for two weeks starting the day after surgery) plus an antibiotic and steroid eye drop association (QID for the first week and BID for the second week) will be given concurrently to 31 patients.
  Interventions: Drug: Dexamethasone+Tobramycin eye drop; Drug: Bromfenac eye drop

INTERVENTIONS:
Drug: Dexamethasone+Tobramycin eye drop — dexamethasone 0.1% and tobramycin 0.3% ophthalmic suspension
Drug: Bromfenac eye drop — bromfenac ophthalmic solution 0.09%
  Other Names: Yellox
  Arms: Bromfenac

SUMMARY:
OBJECTIVE To evaluate the efficacy of bromfenac ophthalmic solution 0.09% for reducing postoperative inflammation in eyes with pseudoexfoliation syndrome (PEX) undergoing cataract surgery and receiving standard postoperative eye drops (dexamethasone 0.1% plus tobramycin 0.3% ophthalmic solution).

DESIGN Two arms, parallel group, randomized, single center, prospective, phase IV clinical trial.

PARTICIPANTS Sixty-two subjects with PEX and cataract will be sequentially assigned, according to a computer-generated randomization list (1:1), to bromfenac (n = 31) or not (n = 31).

INTERVENTION Cataract surgery by means of phacoemulsification and implantation of posterior-chamber intraocular lens will be performed by two experienced ophthalmic surgeons.

Standard Arm: only a standard antibiotic and steroid ophthalmic suspension will be given starting the day after the surgery for two weeks, dosed QID for the first week and BID for the second week (dexamethasone 0.1% and tobramycin 0.3% eye drops association).

Experimental Arm: eyes will receive bromfenac BID for two weeks starting the day after surgery. Standard post-operative topical antibiotic and steroid will be also given concurrently, dosed QID for the first week and BID for the second week (dexamethasone 0.1% and tobramycin 0.3% eye drops association).

Measurements will be carried out at baseline and after one day, 3 days, 1 week and 4 weeks from cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

* cataract
* pseudoexfoliation syndrome

Exclusion Criteria:

* history of ocular inflammation or trauma
* previous intraocular surgery
* corneal haze
* retinal vascular disease
* diabetic retinopathy
* variation of the foveal profile at OCT (macular edema, epiretinal membrane)
* moderate to severe age related macular degeneration

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in anterior chamber inflammation measured by Laser Flare Photometry (photon counts per millisecond) | Baseline, Day 3
  Reduction of 30% of anterior chamber inflammation evaluated by Laser Flare Photometry (LFP) in the bromfenac arm when compared to the non-bromfenac arm at postoperative day 3.

SECONDARY OUTCOMES:
Proportion of patients with central macular thickness greater than 300 microns | Baseline, Week 4
  Macular thickness will be evaluated by Spectral Domain Optical Coherence Tomography (SD-OCT).
Proportion of subjects with best corrected visual acuity equal to 20/20 | Baseline, Week 1
Proportion of patients who had no ocular pain | Baseline, Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Marco Coassin, MD PhD, Principal Investigator — Arcispedale S. Maria Nuova IRCCS; Luigi Fontana, MD PhD, Study Chair — Arcispedale S. Maria Nuova IRCCS
Locations (1):
- Arcispedale Santa Maria Nuova IRCSS - Ophthalmology, Reggio Emilia, RE, Italy